CLINICAL TRIAL: NCT05963594
Title: A Randomized, Double-Blind, Comparator-Controlled, Crossover Study to Evaluate the Post-Prandial Metabolic Effects of Oligomalt in Adults With Type 2 Diabetes (T2D) and in Otherwise Healthy Adults With Overweight or Obesity (HAO)
Brief Title: To Evaluate the Post-Prandial Metabolic Effects of Oligomalt in Adults With T2D and in HAO
Acronym: LORIS-02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 22.06.CLI
Record Dates: First submitted 2023-06-21; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Dietary Supplement
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- T2D Sequence AB (Active Comparator): Where A = 50 g Oligomalt and B = 50 g Glucidex 40.
  Interventions: Dietary Supplement: Oligomalt; Dietary Supplement: maltodextrin
- T2D Sequence BA (Active Comparator): Where A = 50 g Oligomalt and B = 50 g Glucidex 40.
  Interventions: Dietary Supplement: Oligomalt; Dietary Supplement: maltodextrin
- HAO Sequence ABCD (Active Comparator): Where A = 50 g Oligomalt, B = 50 g Glucidex 40, C = 33 g Oligomalt, and D = 33 g maltodextrin Glucidex 40.
  Interventions: Dietary Supplement: Oligomalt; Dietary Supplement: maltodextrin
- HAO Sequence BDAC (Active Comparator): Where A = 50 g Oligomalt, B = 50 g Glucidex 40, C = 33 g Oligomalt, and D = 33 g maltodextrin Glucidex 40.
  Interventions: Dietary Supplement: Oligomalt; Dietary Supplement: maltodextrin
- HAO Sequence DCBA (Active Comparator): Where A = 50 g Oligomalt, B = 50 g Glucidex 40, C = 33 g Oligomalt, and D = 33 g maltodextrin Glucidex 40.
  Interventions: Dietary Supplement: Oligomalt; Dietary Supplement: maltodextrin
- HAO Sequence CADB (Active Comparator): Where A = 50 g Oligomalt, B = 50 g Glucidex 40, C = 33 g Oligomalt, and D = 33 g maltodextrin Glucidex 40.
  Interventions: Dietary Supplement: Oligomalt; Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: Oligomalt — The investigational product (Oligomalt) dissolved in 300 ml water will be consumed over approximately 10 minutes in the morning of the study visit after a fasting period of at least 10 hours.
Dietary Supplement: maltodextrin — The investigational product (maltodextrin) dissolved in 300 ml water will be consumed over approximately 10 minutes in the morning of the study visit after a fasting period of at least 10 hours.
  Other Names: Glucidex 40

SUMMARY:
The goal of this mechanistic, exploratory study is to compare the effectiveness of Oligomalt to Glucidex 40 after eating in adults with Type 2 Diabetes (T2D) and in otherwise healthy adults with overweight or obesity (HAO).

DETAILED DESCRIPTION:
The main question it aims to answer is how consumption of Oligomalt, a slowly digestible carbohydrate, will reduce glucose and insulin spikes in adults with T2D and in HAO relative to Glucidex 40.

ELIGIBILITY:
Type 2 Diabetes (T2D)

Inclusion criteria:

1. Willing and able to sign written informed consent prior to study entry.
2. Male or female, >18 years of age.
3. Established diagnosis of T2D (documented by either HbA1c 6.5 - 10.0% or a history of T2D diagnosis).
4. Treatment naïve or on active therapy with metformin at a daily dose of 1000-3000 mg at screening. Dose of metformin must have been stable for at least 3 months prior to screening.
5. Participants must have a hematocrit value greater than or equal to 34.0% for females and 40% for males.
6. Participants must have a hemoglobin value greater than or equal to 11.0 g/dL for females and 13.5 g/dL for males.

Exclusion Criteria:

1. Type 1 diabetes.
2. Known food allergy or intolerance to study products.
3. Major medical/surgical event in the last 3 months potentially interfering with study procedures and assessments.
4. Abnormal bowel transit, history of a gastrointestinal disorder (e.g., inflammatory bowel disease, diverticular diseases, colon cancer), or history of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average or chronic or recurrent diarrhea with spontaneous bowel movements more often than 3 times daily.
5. Any concomitant medication potentially interfering with study procedures and assessment: such as antibiotics, antiacids, or other medications impacting transit time, colonoscopy, irrigoscopy or other bowel cleansing procedures 4 weeks prior to dosing.
6. Current use of injectable insulin therapy, any other oral (other than metformin) or injectable glucose-lowering drug. Current use of weight loss interventions or treatment with anorectic drugs (e.g., GLP-1 receptor analogues).
7. Current treatment with anticoagulants or antithrombotic agents (warfarin, NOACs, heparin, platelet inhibitors).
8. Current treatment with systemic steroids (application of inhaled or topical steroids is permitted).
9. Recent episode of an acute gastrointestinal illness.
10. Alcohol intake higher than 2 servings per day. A serving is 0.4 dl/1.41 ounces of strong alcohols, 1 dl/3.5 ounces of red or white wine, or 3 dl/10.6 ounces of beer.
11. Current daily cigarette smoking.
12. Are unable to comply with protocol procedures in the opinion of the investigator.
13. Have a hierarchical link with the research team members.
14. Positive pregnancy test or breast-feeding at screening.
15. Participants who have been dosed in another clinical study with any investigational drug/new chemical entity within 30 days or 5 half-lives (whichever is longer) prior to screening.
16. Donation of blood or significant amount of blood loss within 8 weeks prior to screening. Participants must also agree to not donate blood within 8 weeks after their last visit.

HAO:

Otherwise Healthy Adults (HAO) with overweight or obese but who DO NOT present with a confirmed diagnosis of diabetes mellitus

Inclusion criteria:

1. Willing and able to sign written informed consent prior to study entry.
2. Male or female, >18 years of age.
3. BMI ≥ 25 kg/m2.
4. Fasting plasma glucose (FPG) ≤ 125 mg/dL.

Exclusion criteria:

1. Type 1 or type 2 diabetes (including those potentially detected at screening).
2. 2-h plasma glucose ≥ 200 mg/dL - if measured within 6 weeks prior to screening.
3. Known food allergy or intolerance to study products.
4. Major medical/surgical event in the last 3 months potentially interfering with study procedures and assessments.
5. Abnormal bowel transit, history of a gastrointestinal disorder (e.g., inflammatory bowel disease, diverticular diseases, colon cancer), or history of chronic constipation with passage of fewer than 3 spontaneous bowel movements per week on average or chronic or recurrent diarrhea with spontaneous bowel movements more often than 3 times daily.
6. Any concomitant medication potentially interfering with study procedures and assessment: such as antibiotics, antiacids, or other medications impacting transit time, colonoscopy, irrigoscopy or other bowel cleansing procedures four weeks prior to dosing.
7. Current use of injectable insulin therapy, any oral or injectable glucose-lowering drug.
8. Current use of weight loss interventions or treatment with anorectic drugs (e.g., GLP-1 receptor analogues).
9. Current treatment with anticoagulants or antithrombotic agents (warfarin, NOACs, heparin, platelet inhibitors).
10. Current treatment with systemic steroids (application of inhaled or topical steroids is permitted).
11. Recent episode of an acute gastrointestinal illness.
12. Alcohol intake higher than 2 servings per day. A serving is 0.4 dl/1.41 ounces of strong alcohols, 1 dl/3.5 ounces of red or white wine, or 3 dl/10.6 ounces of beer.
13. Current daily cigarette smoking.
14. Are unable to comply with protocol procedures in the opinion of the investigator.
15. Positive pregnancy test or breast-feeding at screening.
16. Participants who have been dosed in another clinical study with any investigational drug/new chemical entity within 30 days or 5 half-lives (whichever is longer) prior to screening.
17. Donation of blood or significant amount of blood loss within 8 weeks prior to screening. Participants must also agree to not donate blood within 8 weeks after their last visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve (iAUC) of post-prandial glycemic excursion induced by Oligomalt relative to maltodextrin over the observation period: iAUC 0-1 hour, iAUC 0-2 hours, iAUC 0-3 hours. | Over the course of 3 hours following study product intake
  Comparisons in the T2D group: 50 g Oligomalt vs 50 g Glucidex 40. Comparisons in the HAO group: 33 g Oligomalt vs 33 g Glucidex 40 and 50 g Oligomalt vs 50 g Glucidex 40.

SECONDARY OUTCOMES:
Total blood glucose AUC | Over the course of 3 hours following study product intake
Blood glucose (iCmax) | Over the course of 3 hours following study product intake
  Maximum blood glucose level
Blood glucose (Cmin) | Over the course of 3 hours following study product intake
  Minimum blood glucose level
Blood glucose (Tmax) | Over the course of 3 hours following study product intake
  Time point at which maximum blood glucose level is measured
Blood glucose (Tmin) | Over the course of 3 hours following study product intake
  Time point at which minimum blood glucose level is measured
Number of participants with glucose levels less than or equal to 3.9 mmol/L | Over the course of 3 hours following study product intake
Number of participants with glucose levels less than or equal to 3.1 mmol/L | Over the course of 3 hours following study product intake
Serum insulin level | Over the course of 3 hours following study product intake
Insulinogenic index (IGI) | 30 minutes
  A measure of early β-cell capacity (first- phase insulin response)
Insulin index | Over the course of 2 hours following study product intake
Matsuda Index (MI) | Over the course of 2 hours following study product intake
Plasma glucagon-like peptide 1 (GLP-1) | Over the course of up to 3 hours following study product intake
Plasma peptide tyrosine (PYY) | Over the course of up to 3 hours following study product intake

OTHER OUTCOMES:
Plasma glucose at individual timepoints | Over the course of 3 hours following study product intake
Between-group comparison of changes in glucose slope | From the time point at which maximum glucose level is measured to 3 hours
Between group comparison of mean "Interquartile range" | Over the course of 3 hours following study product intake
  IQR is defined as the difference between mean Q1 and mean Q3 glucose levels (mmol/L)
Serum insulin at individual timepoints | Over the course of 3 hours following study product intake
Plasma glucagon-like peptide 1 (GLP-1) at individual timepoints | Over the course of 2 hours following study product intake
Plasma peptide tyrosine (PYY) at individual timepoints | Over the course of 2 hours following study product intake
Plasma glucagon-like peptide 1 (GLP-1) | Over the course of 1 hour following study product intake
Plasma peptide tyrosine (PYY) | Over the course of 1 hour following study product intake

CONTACTS AND LOCATIONS:
Overall Officials: Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (1):
- Orange County Research Center, Tustin, California, United States

IPD SHARING:
Plan to Share IPD: No